CLINICAL TRIAL: NCT00794924
Title: Effects of Commercially Available Probiotics on Hospital Outcome
Brief Title: Probiotics and Hospital Outcome in the Elderly
Acronym: PROAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaplan-Harzfeld Medical Center (Other)
Responsible Party: Hilla Zharoni, Chief dietician, Harzfeld Geriatric Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Probiotics and elderly
Record Dates: First submitted 2008-10-28; First posted 2008-11-20 (Estimated); Results first posted 2008-11-20 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2008-11

CONDITIONS: Diarrhea; Constipation
Keywords: probiotics; elderly; motility; diarrhea
MeSH Terms: conditions — Diarrhea; Constipation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics, VSL#3 (Experimental): Acutely hospitalized elderly patients in a geriatric orthopedic rehabilitation department received commercially available probiotics (VSL#3) for 45 days.
  Interventions: Dietary Supplement: VSL#3
- Placebo (Placebo Comparator): Acutely hospitalized elderly patients in a geriatric orthopedic rehabilitation department received placebo sachets for 45 days.
  Interventions: Dietary Supplement: VSL#3; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: VSL#3 — one sachet per day, for 45 consecutive days
  Other Names: probiotics; VSL phrma,USA
Dietary Supplement: placebo — one sachet per day, for 45 consecutive days
  Arms: Placebo

SUMMARY:
Probiotics have been shown to reduce the rate of diarrhea and constipation. The purpose of this study was to investigate if probiotics could improve outcome of hospitalized orthopedic elderly patients.

DETAILED DESCRIPTION:
The patients were divided into two groups. One received probiotics for 45 days and the second received placebo. The patients had a clinical and epidemiological as well as nutritional assessment. They were followed-up as for their bowel movements, abdominal pain and nosocomial infections and for the incidence of helicobacter pylori and clostridiume difficille diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were hospitalized in the Department of Geriatric Orthopedic Rehabilitation a week before their enrollment in the study and signed an informed consent.

Exclusion Criteria:

* Known or suspected allergy to any probiotics
* Neutropenia
* Inability to sign an informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2004-02; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilla Zahroni, MA, Principal Investigator — Chief dietician

REFERENCES:
- [Derived] Zaharoni H, Rimon E, Vardi H, Friger M, Bolotin A, Shahar DR. Probiotics improve bowel movements in hospitalized elderly patients--the PROAGE study. J Nutr Health Aging. 2011 Mar;15(3):215-20. doi: 10.1007/s12603-010-0323-3. PMID 21369670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: February 2004 to january 2005, all patients admitted to the Geriatric Rehabilitation Department of the Harzfeld Geriatric Mdical Center
Groups:
- Probiotics: Acutely hospitalized elderly patients in a geriatric orthopedic rehabilitation department received commercially available probiotics (VSL#3) for 45 days.
Period: Overall Study
Arm/Group | Probiotics | Placebo
Started | 174 (14 patients refused to start the study) | 171 (14 patients refused to start the study)
Completed | 114 | 101
Not Completed | 60 | 70
Not completed — Lost to Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 48 | 60
Not completed — Adverse Event | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotics | Placebo | Total
Number analyzed (Participants) | 174 | 171 | 345
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 169 | 165 | 334
Age Continuous [Mean (Standard Deviation); unit: years] | 76.4 (8.5) | 75.7 (8.6) | 76.05 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 80 | 170
  Male | 84 | 91 | 175

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Number of Days of Either Constipation or Diarrhea in Comparison to the Control Group
Description: Gastrointestinal motility was assessed by the number of days a patient was constipated or had diarrhea.
Time Frame: 45 days of measuring the outcome
Population: The number of participants was chosen in order to receive a difference by GEE statistical model with > 0.05 p value. The analysis was done per protocol.
Measure: Mean (Standard Deviation); unit: days of constipation or diarrhea
Arm/Group | Probiotics | Placebo
Number analyzed (Participants) | 114 | 101
days of constipation or diarrhea | 12 (2.4) | 19 (3.9)

2. Secondary Outcome: Improvement in Nutritional and Immunological Measurements
Time Frame: 45 days
Reporting Status: Not Posted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No